CLINICAL TRIAL: NCT01126047
Title: Validation of Exhaled Carbon Monoxide for DLCO Correction
Brief Title: Exhaled Carbon Monoxide (eCO) for Diffusing Capacity (DLCO) Correction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Eric Kleerup, Clinical Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: eCO
Record Dates: First submitted 2010-05-14; First posted 2010-05-19 (Estimated); Last update posted 2011-11-09 (Estimated); Status verified 2011-11

CONDITIONS: Lung Diseases
Keywords: Lung Diseases
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PFT's, eCO, and pulse oximetry (Other): All subjects in the study will undergo complete pulmonary function testing (spirometry, blood collection for carboxyhemoglobin, diffusing capacity); exhaled carbon-monoxide testing, and pulse oximetry.
  Interventions: Other: eCO testing

INTERVENTIONS:
Other: eCO testing — exhaled carbon monoxide testing measured in duplicate on each of 2 machines immediately prior to the carboxyhemoglobin blood draw and four minutes after the clinical measurement of DLCO

SUMMARY:
The purpose of this study is to check the accuracy of a procedure called exhaled carbon monoxide (eCO) testing. Exhaled carbon monoxide is used by physicians to help assess breathing in people with conditions like asthma and emphysema. eCO may be used to correct another breathing test (called diffusing capacity, or DLCO). Blood collection is usually required to correct the DLCO, so validation of the eCO test may help avoid that blood collection.

DETAILED DESCRIPTION:
The purpose of this study is to check the accuracy of a procedure called exhaled carbon monoxide (eCO) testing. Exhaled carbon monoxide is used by physicians to help assess breathing in people with conditions like asthma and emphysema. 100 subjects who are at least 18 years of age will be invited to participate. The first 50 subjects (Part 1) must have had pulmonary function testing (spirometry, diffusing capacity and CO-oximetry) for clinical reasons ordered by their own physician in order to enroll. The second 50 subjects (Part 2) may undergo this testing as part of the study. Participation requires 1 visit, during which subjects will undergo breathing tests, have blood collected, and answer 3 questions. The number of breathing tests will depend on which part of the study subjects are in. Subjects participating in Part 1 of the study will undergo 2-4 additional diffusing capacity (breathing) tests. (Clinical tests require 2-4 tests. This study requires 6. The number of research tests done depends on the number of clinical tests done. Subjects participating in Part 2 of the study who have not had clinical breathing tests ordered by their physician will undergo 1 spirometry (breathing) test (3-8 blows into a tube), 6 diffusing capacity (breathing tests), and blood draw. All subjects will undergo eCO testing (blowing into a machine) before the breathing tests and after the breathing tests. The visit in Part 1 of the study will take about 30 minutes. The visit in Part 2 of the study will take about 30 minutes for subjects who have undergone clinical breathing tests recently, and about 1 ½ hours for those who must undergo breathing tests for the research. Subjects will also have their pulse oximetry (using a standard finger clip) performed at the same time as each eCO testing.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will at minimum have spirometry, diffusing capacity and CO-oximetry performed for any clinical indication (Part 1 only)
* Willingness to under go the study procedures.
* Ability to give written informed consent to participate in the study.

Exclusion Criteria:

* Subjects on oxygen therapy within 1 hour. High levels of oxygen are used to displace CO in cases of toxicity. Presumably those recently on lower flows of oxygen are not in a steady state for several half-lives.
* Self-reported smoking within 1-hour.
* Significant exercise within 15 minutes
* Recent (within 2 hrs) alcohol consumption (alcohol can interfere with the DLCO measurement)
* Subjects unwilling to remove nail polish from one finger
* Known atypical hemoglobin types (e.g. sickle cell trait or disease, thalassemia etc). The binding and release of oxygen and presumably CO is altered in these types of hemoglobinopathies
* History of known or suspected alveolar hemorrhage. Free hemoglobin or red cells in the alveolus markedly raise the DLCO and theoretically might alter the eCO.
* Known or suspected intestinal bacterial overgrowth. Although the cross reactivity of the CO sensor for hydrogen is <2%, high values of hydrogen from bacterial overgrowth, may lead to erroneous CO measurements.
* Tracheostomy or inability to form a tight seal around the mouthpiece.
* Prior participation in the same part of this study (i.e., subjects can participate in Part 1 and Part 2, but not twice in Part 1, or twice in Part 2)
* Inability to perform spirometry and diffusing capacity
* Inability to consent
* Other diseases or conditions that may, in the opinion of the investigator, result in invalid pulmonary function tests or eCO measurement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-05; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Exhaled carbon monoxide as a predictor of carboxyhemoglobin | 1 year
  Exhaled carbon monoxide will be evaluated as a predictor of carboxyhemoglobin and change in diffusing capacity with increasing carboxyhemoglobin

CONTACTS AND LOCATIONS:
Overall Officials: Michelle R Zeidler, MD, Principal Investigator — UCLA, VA
Locations (2):
- United States (2):
  - UCLA, Los Angeles, California
  - West LA VA, Los Angeles, California